CLINICAL TRIAL: NCT06103461
Title: Fat Grafting an Ideal Filler For Contour Deformities With Hyperpigmentation On Face
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King Edward Medical University (Other)
Responsible Party: Principal Investigator, Afzaal Bajwa, Assistant Professor, King Edward Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: kemu/23/1
Record Dates: First submitted 2023-10-21; First posted 2023-10-26 (Actual); Last update posted 2023-10-26 (Actual); Status verified 2023-10

CONDITIONS: Hyperpigmentation
Keywords: Pigmentation; Contour defect; Fat grafting
MeSH Terms: conditions — Hyperpigmentation

STUDY DESIGN:
Intervention Model Description: Cohort study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Fat Grafting (Experimental): It is an experimental study for effect of fat grafting on pigmentation of skin
  Interventions: Procedure: Autologous fat grafting

INTERVENTIONS:
Procedure: Autologous fat grafting — Autologous fat grafted at contour defects with pigmentary changes

SUMMARY:
Pigmentary changes are commonly associated with contour defects of facial region. These deformities cause cosmetic concerns. Traditionally used techniques indwelling limitations and therefore it invokes innovative techniques to treat contour abrasion and pigmentation simultaneously. The current study focuses on evaluation of the role of autologous fat in improving contour defects of face associated with hyperpigmentation. 100 subjects having contour defects related skin pigmentation were recruited from Feb 2022 till Feb 2023. Fat was harvested, processed under sterilized conditions and grafted into the affected regions of face. The patients were kept under follow up for one year after fat injection. Subjective as well as objective evaluation was done before treatment and one year after fat injection. Results showed significant improvement in pigmentation after fat injection. Most of the patients had high satisfaction regarding improvement in pigmentation and pliability of the grafted area after use of fat graft. A software Image J was applied to objectively showing changes in hyperpigmentation of face after fat graft. In conclusion, utility of autologous fat has effective and promising role as an ideal filler for treating contour defects of face with pigmentary changes

DETAILED DESCRIPTION:
Introduction Facial contour defects need augmentation have pigmentary issues related to them. Such defects are noticed after trauma, autoimmune disease or after infection. These combined contour and pigmentary defects cause social as well as aesthetic concerns. Discolored skin makes them more prominent. Conventionally, fillers are employed but these are short lived at one hand while do not treat pigmentation on the other hand. Body tissues in the form of flaps have also been tried but with the same outcome as with the fillers. Lasers and chemical depigmentation improve skin color but has to do nothing with filling of the contour. In short so far, no single satisfactory remedy is available for such issues. Therefore, some innovative strategy is needed which can fill contour defect and resolves pigmentation too.

Adipose tissue, being autologous, is a pronounced source with regenerative potential as well as natural augmentation. Due to its abundance, easy harvesting and pliability at recipient site make it ideal. Filling effect is just one aspect rather grafted fat not only softens scars, rejuvenates skin but also improves pigmentation. Therefore, in our study we aimed at the evaluation of fat as an ideal filler.

Materials and Methods This prospective study was conducted in Plastic & Reconstructive Surgery Department of KEMU Lahore from Feb 2022 to Feb 2023. Hundred patients of both genders and age between 10 to 50 years having contour defects on face were recruited.

Patients having rejuvenation procedure like filler, laser, depigmentation or PRP done were excluded from the study. Biodata along with deformity details were noted. Advantages, limitations and likely complications related to the procedure were explained and informed consent was documented.

Pre-procedure skin texture, color and defect was noted. Donor area was marked and local anesthesia with 0.5% Xylocain and 1:500,000 Adrenaline in normal saline was infiltrated with one milliliter of fluid for one milliliter of fat to be procured. Fat was procured with blunt 2-mm multi-hole cannula using 10cc Luer-Lok syringe under manual suction applied not more than 2ml. Then fat was transferred to recipient area by using Icc syringe and infiltration canula till symmetry achieved with contralateral respective area of face. Grafted area photographed and integrated color density (ICD1) was found with ImageJ. All patients were observed for 24 hours to look for any complication. Oral analgesic and antibiotics were prescribed for 3 days. Patients were kept under monthly follow up and sessions were repeated if required (13). Subjective as well as objective measurement of outcomes was done. For objective evaluation, repeat photograph was taken after one year of deformity got resolved. Integrated color density (ICD2) was again measured and compared with ICD1. For subjective evaluation, patient's was noted.

Findings were recorded and variables like age, gender, area involved, duration, ICD and satisfaction documented. SPSS 22 used for data analysis with p- Value <0.05 considered significant.

ELIGIBILITY:
Inclusion Criteria:

* Pigmentation with contour defect

Exclusion Criteria:

* Unfit for anesthesia

Ages: 10 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 100 (Actual)
Dates: Start 2022-02-22 (Actual); Primary Completion 2023-02-21 (Actual); Study Completion 2023-02-21 (Actual)

PRIMARY OUTCOMES:
IDC | 6 Months
  integrated color density

CONTACTS AND LOCATIONS:
Overall Officials: Afzaal Bashir, FACS, MS, Principal Investigator — King Edward Medical University, Lahore, Pakistan
Locations (1):
- King Edward Medical University, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No
Statistical data to be shared